CLINICAL TRIAL: NCT00350792
Title: A Phase II Trial Pemetrexed Carboplatin as First Line Chemotherapy for Advanced Non-Small Cell Lung Cancer (NSCLC) in Elderly Patients
Brief Title: Pemetrexed/Carboplatin Non-Small Cell Lung Cancer (NSCLC) Elderly Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9941; H3E-FP-S099 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Results first posted 2009-12-09 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed + Carboplatin (Experimental): Pemetrexed: 500 milligrams per square meter (mg/m^2), intravenous (IV), every 21 days x 6 cycles.
  Carboplatin: Area Under the Curve (AUC) 5, intravenous (IV), every 21 days x 6 cycles.
  Interventions: Drug: pemetrexed; Drug: carboplatin

INTERVENTIONS:
Drug: pemetrexed — 500 milligrams per square meter (mg/m^2), intravenous (IV), every 21 days x 6 cycles
  Other Names: LY231514; Alimta
Drug: carboplatin — Area Under the Curve (AUC) 5, intravenous (IV), every 21 days x 6 cycles

SUMMARY:
A phase II study to evaluate the efficacy and safety profile of the combination of Pemetrexed and Carboplatin in elderly patients with advanced non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Non Small Cell Lung Cancer Stage IIIb (not amenable to radiotherapy treatment) or Stage IV
* No previous chemotherapy for lung cancer
* Men and women > or = 70 years
* At least one uni-dimensionally measurable lesion (Response Evaluation Criteria In Solid Tumors [RECIST]criteria)
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1

Exclusion Criteria:

* Treatment within the last 30 days with a drug that has not received regulatory approval
* Serious systemic disorders
* Inability to discontinue administration of aspirin or anti-inflammatory non steroid
* Concurrent administration of any other antitumor therapy
* Brain metastasis

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-08; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- France (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bobigny
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Le Mans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vandœuvre-lès-Nancy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed + Carboplatin
Started | 62
Completed | 29
Not Completed | 33
Not completed — Adverse Event | 11
Not completed — Death from Study Disease | 1
Not completed — Death from Study Drug Toxicity | 1
Not completed — Death Not Study Drug Related | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 2
Not completed — Lack of Efficacy | 11

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 62
Age Continuous [Mean (Standard Deviation); unit: years] | 76.5 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 51
Region of Enrollment [Number; unit: participants]
  France | 62
Disease Stage [Number; unit: participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body).
  participants
    Stage IIIB | 13
    Stage IV | 49
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 10
    1 - Ambulatory, Restricted Strenuous Activity | 52
Pathological Diagnosis [Number; unit: participants]
  Large Cell Lung Cancer | 5
  Adenocarcinoma of Lung | 32
  Squamous Cell Carcinoma of Lung | 21
  Other: Carcinoma-Infiltrant Indifferencie | 1
  Other: Carcinoma | 1
  Other: Indifferencied Non-Small Cell Lung Cancer | 1
  Other: Undifferentiated | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Complete or Partial Tumor Response (Overall Tumor Response)
Description: Tumor response is defined as the percentage of patients with either a complete response or a partial response. Response was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions and Partial Response=30% decrease in sum of longest diameter of target lesions.
Time Frame: baseline to measured objective tumor response (up to six 21-day cycles)
Population: Patients qualified for tumor response analysis: treated patients, with measurable advanced non-small cell lung cancer (NSCLC) disease and at least one tumor assessment after the patient received at least a first cycle of chemotherapy (unless early progression occurs, including early clinical progressions confirmed by the assessment committee).
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 49
percentage of participants | 28.6 [16.58 to 43.26]

2. Other Pre Specified Outcome: Time to Treatment Failure
Description: Defined as the time from study enrollment to the first observation of disease progression, death as a result of any cause, or early discontinuation of treatment. Time to treatment failure was censored at the date of the last follow-up visit for patients who did not discontinue early, who were still alive, and who have not progressed.
Time Frame: baseline to stopping treatment (up to six 21-day cycles)
Population: All treated patients. 29 patients were censored.
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 62
weeks | 12.95 (0.74)

3. Secondary Outcome: Time to Treatment Failure
Description: as for outcome 2
Time Frame: baseline to stopping treatment (up to six 21-day cycles)
Population: All treated patients. 29 patients were censored.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 62
weeks | 16.0 [10.1 to NA] — Confidence interval is not calculable for the upper limit due to the immaturity of the data.

4. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death. For patients who are alive, overall survival is censored at the last contact.
Time Frame: baseline to date of death from any cause (up to 14.5 months)
Population: Twenty patients were censored as they were still alive at the time of the data cut-off.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 62
months | 10.4 [9.1 to 12.9]

5. Secondary Outcome: Estimated Probability of One Year Progression-free Survival
Description: Progression free survival (PFS) is the duration from enrollment until first disease progression or death. For patients not known to have died as of the data cut-off date and who do not have progressive disease, PFS is censored at the last radiological assessment date.
Time Frame: baseline to measured progressive disease or death, 1 year
Population: Six patients were censored as they had not experienced a qualifying event (death or first disease progression) at the time of data cut-off.
Measure: Median (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pemetrexed + Carboplatin
Number analyzed (Participants) | 62
percentage of patients | 13.1 [4.6 to 21.6]

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Carboplatin
Serious Adverse Events (participants affected / at risk) | 26/62
Other Adverse Events (participants affected / at risk) | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin (N=62)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (6)
Arrhythmia (Cardiac disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Sigmoiditis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 4 (4)
Mucosal inflammation (General disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin (N=62)
Anaemia (Blood and lymphatic system disorders) | 35 (43)
Leukopenia (Blood and lymphatic system disorders) | 12 (23)
Neutropenia (Blood and lymphatic system disorders) | 44 (115)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (68)
Constipation (Gastrointestinal disorders) | 21 (26)
Diarrhoea (Gastrointestinal disorders) | 12 (14)
Nausea (Gastrointestinal disorders) | 21 (32)
Stomatitis (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 14 (17)
Asthenia (General disorders) | 42 (63)
Chest pain (General disorders) | 7 (7)
Oedema peripheral (General disorders) | 5 (5)
Pyrexia (General disorders) | 6 (12)
Weight decreased (Investigations) | 23 (24)
Weight increased (Investigations) | 4 (4)
White blood cell count decreased (Investigations) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 25 (30)
Insomnia (Psychiatric disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days